CLINICAL TRIAL: NCT03237182
Title: The Individualized M(X) Drug-resistant TB Treatment Strategy Study A Strategy to Improve Treatment Outcomes in Patients With Drug-resistant TB
Brief Title: The Individualized M(X) Drug-resistant TB Treatment Strategy Study
Acronym: InDEX
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: WHO 2022 guidelines for DR-TB treatment are set to change. These guidelines recommend the use of an all-oral short course BPAL regimen.Therefore ongoing implementation of the study is considered futile.
Sponsor: Centre for the AIDS Programme of Research in South Africa (Network)
Responsible Party: Principal Investigator, Dr Nesri Padayatchi, Deputy Director, Centre for the AIDS Programme of Research in South Africa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAP 020
Record Dates: First submitted 2017-07-27; First posted 2017-08-02 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Tuberculosis, Multidrug-Resistant
Keywords: whole genome sequencing;
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Intervention Model Description: Patients randomized to the intervention receive a individualized tuberculosis treatment based on whole genome sequencing and the patients randomized to the control receive the standard of care tuberculosis treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized treatment for drug resistant tuberculosis (Experimental): Patients with drug resistance will have whole genome sequencing performed on the respective positive MGIT sample. An individualized TB treatment regimen will be provided to patients based on the whole genome sequencing results
  Interventions: Drug: Individualized TB treatment with multiple drugs
- Standard treatment regimen for drug resistant tuberculosis (Active Comparator): As per South African Department of Health Standard of Care for the treatment of drug resistant tuberculosis
  Interventions: Drug: Standardized TB treatment with multiple drugs

INTERVENTIONS:
Drug: Individualized TB treatment with multiple drugs — Patients with drug-resistant TB will receive a combination of any of the following drugs based on whole genome sequencing:
  rifampicin, rifabutin, isoniazid, high dose isoniazid, pyrazinamide, ethambutol, levofloxacin, moxifloxacin, ofloxacin, gatifloxacin, amikacin, capreomycin, kanamycin, streptomycin, ethionamide, prothionamide, cycloserine, terizidone, pretomanid, linezolid, sutezolid, clofazimine, bedaquiline, delaminid, para-aminosalicylic acid, imipenem/cilastatin, meropenem, amoxicillin/clavulanate, clarithromycin, azithromycin and thioacetazone
  Arms: Individualized treatment for drug resistant tuberculosis
Drug: Standardized TB treatment with multiple drugs — Patients with drug-resistant TB with receive a combination of any of the following drugs based on South African Department of Health guidelines:
  rifampicin, rifabutin, isoniazid, high dose isoniazid, pyrazinamide, ethambutol, levofloxacin, moxifloxacin, ofloxacin, gatifloxacin, amikacin, capreomycin, kanamycin, streptomycin, ethionamide, prothionamide, cycloserine, terizidone, pretomanid, linezolid, sutezolid, clofazimine, bedaquiline, delaminid, para-aminosalicylic acid, imipenem/cilastatin, meropenem, amoxicillin/clavulanate, clarithromycin, azithromycin and thioacetazone
  Arms: Standard treatment regimen for drug resistant tuberculosis

SUMMARY:
This is a randomized controlled clinical trial comparing treatment success of a gene-derived individualized drug-resistant Tuberculosis regimen to a standard Tuberculosis regimen based on South African National Tuberculosis guidelines.

DETAILED DESCRIPTION:
When drug resistance is detected by molecular methods such as the Xpert MTB/RIF assay, second-line Multi Drug-Resistant (MDR) Tuberculosis treatment is started in the complete absence of detailed resistance information. The diagnosis of Multi Drug-Resistant Tuberculosis is confirmed only on availability of Line Probe Assay (LPA)/Drug Susceptibility Testing (DST) results. Extremely Drug-Resistant (XDR) Tuberculosis is diagnosed by in vitro phenotypic resistance to Rifampicin, Isoniazid, fluoroquinolones and injectable second-line drugs (i.e., amikacin, kanamycin, or capreomycin). Existing culture based Drug Susceptibility Testing provides results after 6-8 weeks. This duration may be further increased by other existing laboratory challenges, such as culture contamination.

Furthermore, initial regimens are often not optimal and sometimes completely ineffective as there is a lack of Drug Susceptibility Testing to support them. More importantly, even optimal regimens are changed due to patient intolerance of the drug's side effects.

Whole Genome Sequencing (WGS) has the advantage of determining the complete Deoxyribonucleic acid (DNA) sequence of an organism's genome at a single time point. Using this technology, genotypic mutations conferring resistance to anti-tuberculosis drugs can be identified. This information will assist in identifying not only potential resistant drugs, but also susceptible drugs and thus enable a more accurate and appropriate choice of regimen. In addition, drugs that will not add value to the treatment outcome, but will increase rates of adverse drug reactions, can be eliminated earlier, improving drug-resistant TB treatment outcomes.

In this proposal, we aim to use Mycobacterium Tuberculosis (MTB) whole genome sequencing prior to the selection of a drug-resistant tuberculosis treatment regimen and thus provide an individualized treatment strategy for drug-resistant tuberculosis. By adopting this method, we hope to improve culture negative survival rates at 6 months post treatment initiation .

This study will include 448 adult patients (age ≥ 18 years) that meet inclusion criteria. Patients referred by provincial satellite facilities with microbiological confirmation of drug-resistant tuberculosis (e.g. Xpert MTB/RIF assay / Line Probe Assay) to King DinuZulu Hospital (KDH) will be recruited. Patients randomized to the control arm will receive standard of care (SOC) treatment. Patients randomized to the intervention arm will be given an individualized treatment regimen based on whole genome sequencing conducted on Mycobacteria Growth Indicator Tube (MGIT) positive sputum samples collected at the screening visit.

ELIGIBILITY:
Inclusion Criteria

* Adults ≥ 18 years of age
* Pulmonary Tuberculosis
* Microbiological confirmation [e.g. GeneXpert Mycobacterium Tuberculosis (MTB) detected and Rifampicin (RIF) resistant and / Line Probe Assay (LPA)] of Multi drug-resistant tuberculosis (MDR-TB) / Pre-Extremely drug-resistant tuberculosis (Pre-XDR-TB) / Extremely drug-resistant tuberculosis (XDR-TB)
* Capacity for providing informed consent
* HIV status - HIV infected and uninfected patients are allowed in the study:

  * Patients already on antiretroviral treatment (ART) will be allowed in the study. The antiretroviral treatment regimen will be evaluated for any contraindications to the drugs used.
  * HIV infected patients at any CD4 count irrespective of antiretroviral treatment commencement and duration will be included in the study

Exclusion Criteria:

* Persons suffering from any serious acute condition.
* Any other chronic or clinically significant medical condition that in the opinion of the attending clinician would render the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Culture negative survival rate | 24 months
  To determine if a gene-derived individualized treatment approach in patients with drug-resistant TB will improve culture negative survival rates at 6 months post treatment initiation
Culture negative survival rate | 30 months
  To determine if a gene-derived individualized treatment approach in patients with drug-resistant TB will improve culture negative survival rates at 6 months post treatment initiation

SECONDARY OUTCOMES:
Tuberculosis treatment outcomes | 30 months
  Treatment outcomes are based on treatment success (cure rates and completion of treatment) or mortality or retention in care or time to culture conversion
Rates of adverse events | 30 months
  Rates of adverse events will be compared between arms
Characterization of multi drug-resistant tuberculosis strains | 30 months
  The minimum inhibitory concentrations of Mtb isolates will be correlated with the genotypic mutations detected and the evolution of drug resistance will be monitored by comparing serial isolates from patients
Drug Concentration | 30 months
  To determine the drug concentrations and long-term drug exposures to DR-TB drug regimens in DBS and hair samples respectively
Measure of adherence | 30 months
  To compare adherence to DR-TB drugs using drug concentrations in DBS samples, hair samples, pill count data and participant self-report
Evolution of HIV drug resistance | 30 months
  To assess the evolution of HIV drug resistance in patients receiving Bedaquiline and ART for HIV/MDR-TB treatment
Improved assessment and management of DR-TB | 30 months
  Development of an optimized method for extraction of MTB DNA directly from sputum samples for WGS, compare resistance mutations detected by WGS to current Xpert and LPA; to design a clinical decision-making algorithm for assessment and management of detected resistance mutations

CONTACTS AND LOCATIONS:
Overall Officials: Nesri Padayatchi, MBChB, PhD, Principal Investigator — Centre for the AIDS Programme of Research in South Africa
Locations (1):
- King Dinuzulu Hospital, Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results of the objectives of the study, after deidentification
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Investigators wishing to access data from this study will need to contact the PI to request the data. Requests may be submitted up to 36 months following article publication. Investigators will need to complete a proposal for how the data will be used. The proposal will be reviewed by the CAPRISA Scientific Review Committee and the CAPRISA Executive Committee.

REFERENCES:
- [Background] Musser JM. Antimicrobial agent resistance in mycobacteria: molecular genetic insights. Clin Microbiol Rev. 1995 Oct;8(4):496-514. doi: 10.1128/CMR.8.4.496. PMID 8665467
- [Background] Outhred AC, Jelfs P, Suliman B, Hill-Cawthorne GA, Crawford AB, Marais BJ, Sintchenko V. Added value of whole-genome sequencing for management of highly drug-resistant TB. J Antimicrob Chemother. 2015 Apr;70(4):1198-202. doi: 10.1093/jac/dku508. Epub 2014 Dec 9. PMID 25492392
- [Derived] Maseko TG, Ngubane S, Letsoalo M, Rambaran S, Archary D, Samsunder N, Perumal R, Chinappa S, Padayatchi N, Naidoo K, Sivro A. Higher plasma interleukin - 6 levels are associated with lung cavitation in drug-resistant tuberculosis. BMC Immunol. 2023 Aug 31;24(1):26. doi: 10.1186/s12865-023-00563-2. PMID 37653422